CLINICAL TRIAL: NCT03093337
Title: Early Post Hospital Discharge Psychomotor Therapy Intervention Program: Effect on the Development in Very Preterm Infants at 2-years Corrected Age
Brief Title: Psychomotor Therapy for Very Premature Infants
Acronym: VPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07 227 01
Record Dates: First submitted 2017-03-14; First posted 2017-03-28 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Premature Infant
Keywords: Neuromotor sequelae; Cognitive disorders; Cerebral development; Psychomotoricity; Postural management; Motor coordination; Parenthood
MeSH Terms: conditions — Premature Birth; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychomotor therapy (Experimental): Early post hospital discharge psychomotor therapy.
  Interventions: Other: Early post hospital discharge psychomotor therapy
- Control (No Intervention): No specific support.

INTERVENTIONS:
Other: Early post hospital discharge psychomotor therapy — The intervention consisted on 20 psychomotor therapy sessions between 2 and 9 months, in order to support infants' development, and parent-infant interactions and adjustment. The therapy was based on body and emotional positive feelings and experiences, leading to improve sensory motor and perceptive integration, interactive and exploratory behaviors, physiological and tonic-emotional self-regulation, motor organization and early coordination. The intervention was a partnership with the parents, leading to decode the baby needs and expectations, for the parents to experiment more positive feelings, to become more confident in their own skills and more sensitive, and in synchrony with their baby. Intervention was supported by a detailed assessment scale implemented in the regional network related to the follow-up for vulnerable babies.
  Arms: Psychomotor therapy

SUMMARY:
Our current reflexion is that sensory dys-stimulations, including vestibule-proprioceptive disorders and unbalanced between brain and brainstem maturation of the neonatal period involve an early deviant development for immature infants that will be cascaded through the brain scaffolding and later development. The primary purpose is to determine whether the Early Psychomotor Therapy Intervention Program improves development and behavior in very preterm infants (VPI) at 24-month corrected age (CA).

DETAILED DESCRIPTION:
VPI < 30 week of amenorrhea were randomized, in a simple blind controlled trial. The psychomotor development was evaluated according to the Bayley Scales of Infant Development-III (BSID-III) at 2 years CA. An intermediate point was provided at 9 months CA. Pediatric standardized assessments and psychologist semi-directive interviews were conducted. Parents also completed a self-administering questionnaire relating to the post-traumatic stress. The intervention consisted on 20 therapy sessions between 2 and 9 months CA, in order to support infants' development, and parent-infant interactions and adjustment.

Extended description of the protocol, including more technical information (as compared to the Brief Summary) if desired. Do not include the entire protocol; do not duplicate information recorded in other data elements, such as eligibility criteria or outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Infants with a gestational age between 24 and 30 weeks.

Exclusion Criteria:

* Infants with congenital disease,
* Infants with brain bleeding grade III-IV,
* Infants with periventricular leucomalacia,
* Infants whose mothers had a documented history of physical or mental illness, or drug abuse
* Infants from non-French -speaking families.

Ages: 24 Weeks to 30 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 162 (Actual)
Dates: Start 2007-12-01 (Actual); Primary Completion 2013-12-01 (Actual); Study Completion 2017-07-08 (Actual)

PRIMARY OUTCOMES:
Psychomotor development assessment. | Year 2
  Assessed by the Bayley Scale Third Edition BSID-III.

SECONDARY OUTCOMES:
The acceptability of the protocol by the parents for the intervention group. | Month 9
  Assessed by a self-questionnaire given by the neonatologist at the end of the treatment.
The quality of parenting. | Month 9; Year 2
  Assessed by a grid (established by the team of child psychiatry neonatology).
The clinical evolution of the child assessed by a standardized neurological examination. | Months 3, 6, 9, 12, 18, 24
  Assessed during the consultations planned in the network (neonatologists of the CHU), based on a standardized neurological examination.

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Alberge, MD, Principal Investigator — Hôpital des enfants, Toulouse
Locations (10):
- France (10):
  - CH Albi, Albi, Midi-Pyrénées
  - CH Auch, Auch, Midi-Pyrénées
  - CH Cahors, Cahors, Midi-Pyrénées
  - CH Castres, Castres, Midi-Pyrénées
  - CHIVA centre hospitalier du val d'Ariège, Foix, Midi-Pyrénées
  - CH Montauban, Montauban, Midi-Pyrénées
  - CH Tarbes, Tarbes, Midi-Pyrénées
  - Hôpital des enfants, Toulouse, Midi-Pyrénées
  - Clinique Sarrus Teinturiers, Toulouse, Midi-Pyrénées
  - Clinique Ambroise Paré, Toulouse, Midi-Pyrénées

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shevell MI, Bodensteiner JB. Cerebral palsy: defining the problem. Semin Pediatr Neurol. 2004 Mar;11(1):2-4. doi: 10.1016/j.spen.2004.01.001. PMID 15132247
- [Background] Hagberg B, Hagberg G, Beckung E, Uvebrant P. Changing panorama of cerebral palsy in Sweden. VIII. Prevalence and origin in the birth year period 1991-94. Acta Paediatr. 2001 Mar;90(3):271-7. PMID 11332166
- [Background] Nelson KB. Can we prevent cerebral palsy? N Engl J Med. 2003 Oct 30;349(18):1765-9. doi: 10.1056/NEJMsb035364. No abstract available. PMID 14585946
- [Background] Jacobsson B, Hagberg G. Antenatal risk factors for cerebral palsy. Best Pract Res Clin Obstet Gynaecol. 2004 Jun;18(3):425-36. doi: 10.1016/j.bpobgyn.2004.02.011. PMID 15183137
- [Background] Palisano R, Rosenbaum P, Walter S, Russell D, Wood E, Galuppi B. Development and reliability of a system to classify gross motor function in children with cerebral palsy. Dev Med Child Neurol. 1997 Apr;39(4):214-23. doi: 10.1111/j.1469-8749.1997.tb07414.x. PMID 9183258
- [Background] Weisglas-Kuperus N, Koot HM, Baerts W, Fetter WP, Sauer PJ. Behaviour problems of very low-birthweight children. Dev Med Child Neurol. 1993 May;35(5):406-16. PMID 7684346
- [Result] Alberge C, Ehlinger V, Noack N, Bolzoni C, Colombie B, Breinig S, Dicky O, Delobel M, Arnaud C. Early psychomotor therapy in very preterm infants does not improve Bayley-III scales at 2 years. Acta Paediatr. 2023 Sep;112(9):1916-1925. doi: 10.1111/apa.16848. Epub 2023 Jun 5. PMID 37191836